CLINICAL TRIAL: NCT05409313
Title: Tailored Training Empowers Hospital Nurses' Competency and Application of Evidence-based Practice and Shared Decision-making: a Randomized Controlled Trial
Brief Title: EBP-SDM Training Program Empowers Nurses' Competency and Performance
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Cheng-Hsin General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: CHGH110-IU09
Record Dates: First submitted 2022-02-20; First posted 2022-06-08 (Actual); Last update posted 2022-06-08 (Actual); Status verified 2022-06

CONDITIONS: Training; Nurse; Evidence-based Practice

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EBP and SDM training group (Experimental): A total of 36 nurses will be received EBP and SDM training program.
  Interventions: Behavioral: EBP training; Behavioral: SDM training
- SDM training group (Active Comparator): A total of 36 nurses will be received SDM training alone.
  Interventions: Behavioral: SDM training

INTERVENTIONS:
Behavioral: EBP training — The EBP training program was modified by the 5A-steps EBP teaching model that which aimed to enhance nurses' EBP competencies and application. A 12-hours EBP training consisted of lectures, hand-on practice, group and individual consulting, group presentations and reflections, and disseminating findings to publish.
  Arms: EBP and SDM training group
Behavioral: SDM training — A 10-hour SDM training program included lecture 4 hours and workshops 6 hours, with focused on 3-talk model for SDM skills, 4-habit model for communication skill, and how to use Ottawa personal decision guide. Teaching strategies included lectures, clinical scenarios role play, and post-scenario debriefing. The major contents were SDM concepts and essential steps, SDM tools, strategies for the clinical implementation, the concept and purpose of choosing wisely campaign, and patient-centered communication skills.

SUMMARY:
The purpose of this study will be to evaluate the effect on competency and performance of EBP and SDM.

1. To evaluate the effect of the 5As-steps EBP training program on competency in nurses-midwives
2. To evaluate the effect of the SDM training program on performance in in nurses-midwives

DETAILED DESCRIPTION:
This is a randomized controlled trial with repeated measures at four time points which are before the start of the intervention (Baseline), classroom teaching (posttest 1), clinical practice (posttest 2), and follow-up (posttest 3). The experimental group will receive the tailored EBP-SDM training program both in classroom and clinical settings.A total of 72 nurses will be recruited from one hospital.

The interventions of this study will integrate classroom activities with practical learning experiences. The investigators previously developed the teaching model of 5As-steps EBP which will be use as framework for the teaching. Teaching activities involve lectures, group and individual consulting, hand-on activities, clinical cases, role play exercises, and debriefing. Previous researchers described the fundamental principles and the 5 steps of EBP and adapted those principles into their 5As-steps EBP model as shown in the following figure. The first step is asking. Nurses-midwives have to establish a well-built clinical question with all the components facilitating performance literature review for relevant database. Step two is acquiring in which nurse-midwives efficiently find the best relevant evidence to answer the question. The third step is appraising meaning that nurse-midwives carefully and systematically examining the trustworthiness of research findings. The fourth step is applying of the appraised evidence to the patients. This step requires integrating the best evidence with clinical expertise and patients' unique values and preference. The final step assessing the outcomes. At this step, nurse-midwives evaluate effectiveness and efficacy of the performance and change in practice. With conscientious application of these 5 steps, each time the cycle completes a turn, patient care and clinical practice is improved.

The Ottawa Decision Support Framework will be use as framework for the teaching. As shown in the following figure, Ottawa Decision Support Framework summarizes three elements in SDM, which are decisional needs, decision outcomes, and decision support . This framework integrates viewpoints from social psychology, economics and social support, and applies to all individuals taking part in decision making including the patients, family members and healthcare providers.

Instruments is listed as following:

(1)Health Sciences-Evidence Based Practice (HS-EBP);(2)9-item Shared Decision-Making Questionnaire (SDM-Q-9 and SDM-Q-Nr);(3)OPTION5;(4)Four Habits Coding Scheme (4HSC);(5)Brief Decision Support Analysis (DSAT-10);(6)Demographic Questionnaire;(7)SURE Test.

ELIGIBILITY:
Inclusion Criteria:

* Work more than 3 months
* Registered Nursing in Taiwan

Exclusion Criteria:

* Not providing care in clinical.
* On-job and received the school education.
* Received the training program of EBP.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2021-03-31 (Actual); Primary Completion 2024-03-31 (Estimated); Study Completion 2024-03-31 (Estimated)

PRIMARY OUTCOMES:
Participant characteristics questionnaire | before intervention
  The structured questionnaire designed by researcher. Participants' characteristics included age, sex, educational level, working unit, nursing clinical ladder, and nursing specialties. Participants' self-rated EBP-related abilities included English capability, previous evidence-based nursing learning, experiences, and practice.
Change is assessed of Health Sciences-Evidence Based Practice questionnaire | Change from baseline, Week 2, Week 6, and Week 10
  The outcome of EBP competency and application was measured by the Health Sciences-Evidence Based Practice (HS-EBP) questionnaire, which aimed to assess EBP knowledge, attitudes, behavior, skills, as well as barriers and facilitators of EBP (Fernández-Domínguez et al., 2017). The HS-EBP contained 60 items that divided into five domains: beliefs-attitudes (12 items), results from scientific research (14 items), development of professional practice (10 items), assessment of results (12 items), and barriers-facilitators (12 items). A 10-point Likert scale from 1 to 10 was used for each item for measuring the degree of agreement with respect to EBP competency. A higher HS-EBP score indicated the greater the degree of agreement.
Change is assessed of SDM-Q-9 and SDM-Q-Nr questionnaire | Change from baseline, Week 2, Week 6, and Week 10
  The SDM-Q-9 and SDM-Q-Nr were developed for using in adult clinical setting, it has been adapted to address the SDM between healthcare providers and the patient in separate studies resulting in consistent testing (Scholl et al., 2012). Both SDM-Q-9 and SDM-Q-Nr contain nine items with responses on a 6-point Likert scale ranging between "completely disagree" and "completely agree". A total raw score between 0 and 45 was calculated by summing the scores of all items. The total raw score was transformed by the (Raw Score*20)/9 formula to create a sum score ranged between 0 and 100. This process assumes that the extent of SDM is additive, therefore, a higher score represents higher perceived SDM.
Change is assessed of DSAT-10 questionnaire | Change from baseline and Week 10
  The DSAT-10 was used to evaluate the quality of decision support provided by health professionals to patients facing tough health decisions (Stacey et al., 2008). Each item as present "1" or absent "0" within the encounter. This 10-item scale had adequate inter-rater reliability (kappa = 0.55) and agreement for encounters involving trained nurses (kappa = 0.62) (Stacey et al., 2008).
Change is assessed of OPTION5 questionnaire | Change from baseline and Week 10
  OPTION5 is a brief, theoretically grounded observer measure of SDM based on the talk model (Elwyn et al., 2005). The five items of OPTION5 replicated the response format, assessment, and scoring methods of OPTION12. The scale was designed to measure the magnitude of skill. The scale scoring guidance as, the behavior was not observed "0", a minimal attempt was made to exhibit the behavior "1", asked about patient's preference "2", the behavior was exhibited to a good standard "3", and the behavior was observed and executed to a high standard "4". A total score ranged between 0 and 20, and rescaled between 0 and 100. The adequate inter-rater reliability of OPTION5 was presented by the intra-class correlation (ICC = 0.67).
Change is assessed of Four Habits Coding Scheme questionnaire | Change from baseline and Week 10
  The Four Habits Coding Scheme (4HCS) used to assess and quantify clinicians' communication behaviors from an external rater's perspective (Krupat et al., 2006). The 23-item 4HCS derived from the core skills in communication. Each item was rated on a 5-point scale which the midpoint and the two endpoints in specific behavioral terms indicated that the clinician used little or no jargon "1", some jargon "3", and highly technical "5". Rather than focusing on frequency counts of behavior, each item of the 4HCS was rated on five levels of performance on a 5-point Likert scale, ranging from 1 (not very effective) to 5 (high effective). A total score for each dimension can be calculated by summing the scores of all items of that dimension. Higher scores indicated better performance. The reliability of the 4HCS, the inter-rater coefficients ranged between .69 and .80 (Krupat et al., 2006).
Change is assessed of SURE test questionnaire | Change from baseline and Week 10
  The SURE test was based on the Ottawa Decision Support framework to screen for decisional conflict in patients facing clinical decisions in primary care (Légaré et al., 2010). Each item had a response of yes scoring "1" and a response of no scoring "0", with combined total scores from 4 items less than 4 indicating the patient experiencing decisional conflict. The SURE test showed adequate internal consistency of Kuder-Richardson 20 coefficient of 0.7 (Ferron Parayre et al., 2014).

CONTACTS AND LOCATIONS:
Overall Officials: Mei-ling Yeh, Professor, Study Chair — School of Nursing National Taipei University of Nursing and Health Sciences
Locations (1):
- Cheng Hsin General Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No